CLINICAL TRIAL: NCT04935034
Title: Absorption Kinetics and Efficacy of Vitamin D Enriched Supplements in Older Adults.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College Dublin (Other)
Responsible Party: Principal Investigator, Aifric O'Sullivan, Assistant Professor, University College Dublin
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: LS-20-53-OSullivan-McCourt
Record Dates: First submitted 2021-06-15; First posted 2021-06-22 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Vitamin D Deficiency
MeSH Terms: conditions — Vitamin D Deficiency

STUDY DESIGN:
Intervention Model Description: The is a 4 arm single-blinded crossover study
Who Masked: Participant
Masking Description: single-blinded crossover study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Vitamin D enriched mixed micelles dairy drink (Experimental): 20ug vitamin D in pre-formed mixed micelle dairy drink
  Interventions: Dietary Supplement: Vitamin D supplement
- Vitamin D enriched olive oil dairy drink (Active Comparator): 20ug vitamin D in olive oil dairy drink
  Interventions: Dietary Supplement: Vitamin D supplement
- Vitamin D enriched fish oil dairy drink (Active Comparator): 20ug vitamin D in fish oil dairy drink
  Interventions: Dietary Supplement: Vitamin D supplement
- Vitamin D enriched fat-free dairy drink (Active Comparator): 20ug vitamin D in fat-free dairy drink
  Interventions: Dietary Supplement: Vitamin D supplement

INTERVENTIONS:
Dietary Supplement: Vitamin D supplement — This intervention will compare the effect of changing the lipid component of a vitamin D enriched dairy drink on postprandial change in 25OHD concentrations.

SUMMARY:
The proposed study will examine vitamin D bioavailability when 20µg of vitamin D is consumed in 5 different forms:

i) a vitamin D enriched pre-formed mixed micelle dairy drink ii) a vitamin D enriched olive oil dairy drink iii) a vitamin D enriched fish oil dairy drink iv) a vitamin D enriched fat-free dairy drink

DETAILED DESCRIPTION:
This postprandial study will recruit healthy males and females aged 18 and over. Upon completion of informed consent procedures and successful screening, the volunteers will complete 4 study visits. Participants will consume a standardised meal the evening before each test day, and will arrive in the morning to the research facility in UCD after an overnight fast of 12 hours.

On the study test days, volunteers will be given one of the following vitamin D treatments in a dairy drink, followed by a low-fat breakfast.

1. mixed micelles
2. olive oil
3. fish oil
4. fat-free

Participants will also be given a low-fat lunch 5 hours after the supplement is consumed. Volunteers will be cannulated by a trained phlebotomist on arrival, and a fasting blood sample will be taken. Following ingestion of the vitamin D supplements blood samples will be taken at 0,2,4,6, and 8 hours post ingestion. A 10mL sample will be collected at each time point. In total, 60mL of blood will be collected over 24 hours. The participant's food intake will be recorded during the visit.

ELIGIBILITY:
Inclusion Criteria:

Healthy men and women

Exclusion Criteria:

Pregnant or lactating Smokers Individuals that are not free-living e.g. institutes where meals are prepared in bulk such as nursing homes, prisons etc.

An inability to read, write or understand English Following a strict prescribed diet for any reason, insulin dependent diabetes, coeliac disease, Crohn's disease Disease or condition that requires chronic therapeutic nutritional or medical treatment.

Those taking supplemental vitamin D Those who have been on a sun holiday in the last 2 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Change in 25-hydroxyvitamin D (25(OH)D) | 8 hours
  Change in 25(OH)D up to 8 hours after consuming the vitamin D enriched dairy drink

CONTACTS AND LOCATIONS:
Locations (1):
- University College Dublin, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No
At the start of the study each participant will have a study code assigned to them. All of the data from the trials will be stored using these unique study codes. A file will be set up which will be stored in a location separate to the study data. This file will contain a list which will link each participants contact details to the corresponding ID code. All stored information will be encrypted and protected by a password that only the researcher and PI will know.